CLINICAL TRIAL: NCT03772262
Title: Assessing Goldenseal-drug Interactions Using a Probe Drug Cocktail Approach
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Washington State University (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Mary Paine, Professor, Washington State University
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 16620; U54AT008909 (NIH)
Record Dates: First submitted 2018-10-01; First posted 2018-12-11 (Actual); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: Interaction Drug Food
Keywords: Pharmacokinetics; Goldenseal; Metformin; Furosemide; Rosuvastatin; Midazolam; Natural product
MeSH Terms: interventions — Metformin; Furosemide; Midazolam; Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (Experimental): Study subjects will be administered a single dose of midazolam syrup (2.5 mg), metformin solution (50 mg), furosemide solution (1 mg), and one rosuvastatin tablet (10 mg) by mouth. Plasma will be collected from 0-96 hours. Urine will be collected from 0-24 hours.
  Interventions: Drug: Metformin; Drug: Furosemide; Drug: Midazolam oral solution; Drug: Rosuvastatin Oral Tablet
- Treatment (Experimental): Study subjects will be administered goldenseal 2 capsules (500 mg each) three times daily for 5 days. On day 6, subjects will be administered goldenseal 2 capsules (500 mg each), a single dose of midazolam syrup (2.5 mg), metformin solution (50 mg), furosemide solution (1 mg), and one tablet (10 mg) rosuvastatin. Goldenseal 2 capsules (500 mg each) will be administered approximately 4 and 8 hours later. Plasma will be collected from 0-96 hours. Urine will be collected from 0-24 hours.
  Interventions: Dietary Supplement: goldenseal; Drug: Metformin; Drug: Furosemide; Drug: Midazolam oral solution; Drug: Rosuvastatin Oral Tablet

INTERVENTIONS:
Dietary Supplement: goldenseal — Oral 500 mg capsules
  Arms: Treatment
Drug: Metformin — Oral solution
Drug: Furosemide — Oral solution
Drug: Midazolam oral solution — Oral syrup
Drug: Rosuvastatin Oral Tablet — Oral tablet

SUMMARY:
Goldenseal is a botanical natural product commonly used to self-treat symptoms of the common cold and many digestive disorders. Goldenseal products typically contain the isoquinoline alkaloids berberine, hydrastine, and hydrastinine. These constituents contain a methylenedioxyphenyl ring, a 'structural alert' that can lead to irreversible inhibition of drug metabolizing enzymes, particularly the cytochromes P450 (CYPs). Clinical studies involving healthy volunteers demonstrated that, compared to baseline (absence of goldenseal), CYP2D6 and CYP3A activities were reduced by 40-60% following treatment with goldenseal. Compared to the CYPs, the effects of goldenseal products on drug transporters are understudied, particularly in human subjects. Using a 'cocktail' consisting of 'probe' drug substrates for CYP3A and various transporters, the effects of goldenseal on the pharmacokinetics of each probe drug will be examined in healthy volunteers. Results will provide useful information about the risk of co-consuming goldenseal with additional drugs that are substrates for transporters.

DETAILED DESCRIPTION:
Many patient groups often supplement their pharmacotherapeutic regimens with herbal and other natural products (NPs), raising concern for adverse interactions with conventional drugs. Unlike for drug-drug interactions, rigorous guidelines for assessing the risk of NP-drug interactions do not exist. The NIH-funded Center of Excellence for Natural Product-Drug Interaction (NaPDI) Research (U54 AT008909) was created in September, 2015. The mission of the NaPDI Center is to provide leadership in the identification, evaluation, and dissemination of potential clinically significant pharmacokinetic NP-drug interactions. One over-arching goal of the Center is to develop a set of Recommended Approaches to guide researchers in the proper conduct of NP-drug interaction studies. These Recommended Approaches will be based on results generated from a series of Interaction Projects that will include mechanistic human in vitro and clinical studies focused on four carefully selected high priority NPs.

Using a systematic approach, the NaPDI Center selected four high priority NPs as precipitants of NP-drug interactions. One of these NPs is goldenseal, which is typically used to self-treat symptoms of the common cold, as well as numerous digestive disorders, both as a single extract and in combination with other NPs, particularly Echinacea spp. Major constituents of goldenseal include the isoquinoline alkaloids berberine, hydrastine, and hydrastinine. These constituents contain a methylenedioxyphenyl ring, a 'structural alert' that can lead to irreversible inhibition of drug metabolizing enzymes, particularly the cytochromes P450 (CYPs). Indeed, clinical studies involving healthy volunteers demonstrated that, compared to baseline (absence of goldenseal), CYP2D6 and CYP3A activities were reduced by 40-60% following administration of ~1 g of a goldenseal extract three times daily for 14 or 28 days .

Compared to the CYPs, the effects of goldenseal products on drug transporters are understudied, particularly in human subjects. A 'cocktail' consisting of 'probe' drug substrates for CYPs and transporters is an efficient, cost-effective means to examine the effects of a precipitant drug or NP on the pharmacokinetics of multiple object drugs simultaneously. Such cocktails are used frequently by both academia and the pharmaceutical industry to test for the interaction potential of new chemical entities, results of which are often included in drug labels. A number of cocktails exist for the CYPs and have been used successfully over the past 20+ years. A transporter cocktail was described recently that consists of the probe drugs furosemide [organic anion transporter (OAT)1 and OAT3 substrate], metformin [(organic cation transporter 2, multidrug and toxin extrusion protein (MATE)1, and MATE2-K substrate)], and rosuvastatin [organic anion transporting polypeptide (OATP)1B1, OATP1B3, and breast cancer resistance protein substrate].

Based on the multiple scientific gaps with respect to a commonly used NP, the purpose of this healthy volunteer study is to assess the inhibitory effects of a well-characterized goldenseal product on the pharmacokinetics of the aforementioned transporter probe drugs; the CYP3A probe midazolam will be included to serve as a positive control object drug. Results will be used to develop (1) a Recommended Approach regarding clinical study design of NP-drug interactions and (2) mathematical models that can be used to predict the risk of potential goldenseal-precipitated interactions with drugs whose pharmacokinetics are influenced by CYP3A and/or transporters.

ELIGIBILITY:
Inclusion Criteria:

* Ability to participate in the study (time, transportation, etc.)
* Ability to understand the informed consent form
* Men and women aged from 18 to 65 years
* Willingness to abstain from alcohol and caffeinated beverages for the evening prior to and during each in-patient study day
* Willingness to abstain from citrus juices and other dietary supplements for the duration of the study

Exclusion Criteria:

* Any current major illness or chronic illness including but not limited to kidney disease, hepatic disease, diabetes mellitus, hypertension, coronary artery disease, chronic obstructive pulmonary disease, previous stroke or embolic disease history, cancer, and HIV/AIDS
* History of allergy to goldenseal, midazolam, furosemide, metformin, or rosuvastatin
* History of anemia or any other significant hematologic disorder
* History of renal failure or lactic acidosis (metformin)
* History of apnea (midazolam)
* History of heart failure, electrolyte imbalance (furosemide)
* History of hypotension (goldenseal)
* History of drug or alcohol addiction or major psychiatric illness
* Women who are intending to become pregnant within the next three months, are currently pregnant, or are currently breastfeeding
* Out-of-range clinical laboratory value that the study physician considers participation in the study a health risk
* Taking concomitant medications, both prescription and non-prescription (including herbal/natural products) known to alter the pharmacokinetics or pharmacodynamics of midazolam, furosemide, metformin, or rosuvastatin.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2018-04-05 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
midazolam AUC ratio (treatment/control) | 0-96 hours
  ratio of the area under of the plasma concentration time curve (AUC) of midazolam in the presence to absence of goldenseal

SECONDARY OUTCOMES:
midazolam Cmax ratio (treatment/control) | 0-96 hours
  ratio of the maximum plasma concentration (Cmax) of midazolam in the presence to absence of goldenseal

CONTACTS AND LOCATIONS:
Locations (1):
- Washington State University, Spokane, Washington, United States

IPD SHARING:
Plan to Share IPD: No